CLINICAL TRIAL: NCT04505319
Title: Prospective, Single Center Study for the Clinical Evaluation of the Safety and Performance of a Dermal Filler in Correction of Mid-face Age-related Volume Deficit
Brief Title: Clinical Evaluation of the Safety and Performance of a Filler in Correction of Mid-face Age-related Volume Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relife S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReGl/19/Dfc-Res/001
Record Dates: First submitted 2020-07-30; First posted 2020-08-10 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Aesthetics; Intradermal Injections
Keywords: DERMAL FILLER; sodium hyaluronate; RELIFE

STUDY DESIGN:
Intervention Model Description: * prospective,
  * non comparative
  * single centre,
  * on healthy subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEFINISSE CORE FILLER (Experimental): Cross linked sodium hyaluronate 25 mg/ml with 0,3% lidocaine hydrochloride will be inject during the first visit and a touch up after one month if indicated by the physician.
  The filler will inject in the face.
  Interventions: Device: DEFINISSE CORE FILLER

INTERVENTIONS:
Device: DEFINISSE CORE FILLER — DEFINISSE CORE FILLER volume will be injected between 4.0 of 5.0 ml on the whole face (at the discretion of the treating physician to achieve an optimal aesthetic result).
  A touch-up will be possible at the first follow-up visit (after one month) with a amount of product between 4.0 and 5.0 ml on the whole face

SUMMARY:
Prospective, single center study, on healthy subjects to evaluate the aesthetic improvement of facial volume, effect on the restoration and/or augmentation in subjects with mid-face age-related volume deficit after injection of a filler with lidocaine.

DETAILED DESCRIPTION:
Prospective, non comparative, single center study, on healthy female subjects. The scope is to evaluate the performance and safety of a dermal filler (definisse core filler plus lidocaine) to evaluate the aesthetic improvement of facial volume, effect on the restoration and/or augmentation in subjects with mid-face age-related volume deficit after injection of a filler with lidocaine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject;
2. Sex: female;
3. Age: between 40 and 60 years;
4. BMI between 18 and 25 included.
5. Subject having given freely and expressly his informed consent;
6. Subject with a volume deficit on malar area and requiring a correction using a filler;
7. Subject, psychologically able to understand the study related information and to give a written informed consent;
8. Subject affiliated to a health social security system;
9. Female of childbearing potential using a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study and during all the study (oral contraceptives, patch contraceptives, injection contraceptives, male condom with intra-vaginal spermicide, diaphragm or cervical cap with spermicide, vaginal contraceptive ring, intrauterine device, surgical sterilization (bilateral tubal ligation), vasectomized partner, or sexual abstinence).
10. Female subjects of childbearing potential must have a negative pregnancy test at the inclusion;
11. Subject agreeing to keep their usual cleansing / care products on the face during the whole study period;
12. Whole full teething subjects

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Subject in a social or sanitary establishment.
4. Subject participating to another research on human beings or being in an exclusion period for a previous study.
5. Subject having received 4500 euros indemnities for participation in researches involving human beings in the 12 previous months, including participation in the present study.
6. Intensive exposure to sunlight or UV-rays within the previous month and foreseen during the study.
7. Subject with a tattoo, a scar, moles, pigment disorders or anything on the studied zones which may interfere with the study at the investigator appreciation.
8. Subject with unstable weight or planning to do a dietary regime during the study.
9. Subject with too severe mid-face volume deficit.
10. Subjects without teeth or with dental prostheses
11. Subject with severe, ongoing and uncontrolled diseases such as malignancy or history of malignancy, type I diabetes, liver failure, renal failure, lung/heart disease, neoplasia, malignant blood disease, tumor, HIV, epilepsy, porphyria or other major disease, likely to interfere with the measured parameters or to put the subject to an undue risk.
12. Subject with known history of or suffering from autoimmune disease and/or immune deficiency
13. Subject with current cutaneous inflammatory or infectious processes (eg, acne, herpes, mycosis, papilloma, chronic eczema, atopic dermatitis …), abscess, unhealed wound, or a cancerous or precancerous lesion on the studied zone.
14. Subject having history of anaphylactic shock or know allergy or hypersensitivity to hyaluronic acid or to one of the components of the tested device, antiseptic solution, lidocaine hydrochloride or to amide-type local anaesthetics.
15. Subject predisposed to keloids or hypertrophic scarring.
16. Subject with coagulation and/or homeostasis disorders.
17. Subject with a past history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats;
18. Subject having received treatment with a laser, a dermabrasion, a surgery, a chemical peeling, mesotherapy or other ablative procedure on the face within the past 12 months prior to inclusion;
19. Subject having received injection with a reabsorbable filling product in the face area within the past 12 months prior to inclusion;
20. Subject having received at any time injection with a slowly reabsorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of hyaluronic acid (HA) and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …) or with a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …);
21. Subject having received at any time a treatment with suspension threads in the face;
22. Any medication which may interfere, at the interpretation of the investigator, with the study objectives in term of efficacy and safety.
23. Subject under medications which may cause lipoatrophy;
24. Subject using medication such as aspirin, NSAIDs (ibuprofen, naproxen, …), antiplatelet agents, anticoagulants, high-doses vitamin C within 10 days prior to inclusion or being a chronic user;
25. Subject having received chemotherapy agents, immunosuppressive medications or systemic corticosteroids within 3 months of enrolment and during the study.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Global aesthetic improvement one month | one month after injection (first visit from Day 0)
  Clinical evaluation of the global aesthetic improvement (GAIS) one month after injection of the investigational medical device in subjects with mid-face age-related volume deficit.

SECONDARY OUTCOMES:
Global aesthetic improvement during follow up | 3, 6, 9, 12 and 18 months after injection
  Clinical evaluation of the global aesthetic improvement (GAIS) 3, 6, 9, 12 and 18 months after injection of the investigational medical device in subjects with mid-face age-related volume deficit.
Clinical evaluation on restoration and/or augmentation of facial volume | from baseline (Day 0) to 1, 3, 6, 9, 12 and 18 months
  Clinical evaluation of the investigational medical device effect on the restoration and/or augmentation of facial volume, with a clinical scale (FVLS) Face Volume Loss Scale, with a score from Grade 1 to Grade 5, when Grade 1 is the better outcome .
Need of a touch-up injection | after one month of injection (Month 1)
  evaluation if a touch up injection is needed after one month
Objective evaluation on restoration and/or augmentation of facial volume | from baseline (Day 0) to 1, 3, 6, 9, 12 and 18 months
  Objective evaluation of the investigational medical device effect on the restoration and/or augmentation of facial volume, with cheekbone volume variation evaluation by 3D LifeViz® system
subject satisfaction on Aesthetic improvement | at each time point after injection, 1 month, 3 months, 6 months, 9 months, 12 months and 18 months.
  Evaluation of subject satisfaction using a subjective evaluation questionnaire, (GAIS) Global Aesthetic improvement Scale, the scores is from 1 to 5, when 1 is the better outcome.
Evaluation of injector satisfaction on using medical device | During the injection Day 0 and 1 one month after the first injection (Month 1)
  Evaluation of injector satisfaction using a subjective evaluation questionnaire
evaluation on skin quality after injection with Dermascan | from baseline (Day 0) to 3, 6, 9, 12 and 18 months after initial injection
  Objective evaluation of the investigational medical device effect on skin quality using Dermascan instrument
evaluation on skin thickness after injection with Dermascan | from baseline (Day 0) to 3, 6, 9, 12 and 18 months after initial injection
  Objective evaluation of the investigational medical device effect on skin thickness using Dermascan instrument
evaluation onskin biomechanical properties after injection with Cutometer | from baseline (Day 0) to 3, 6, 9, 12 and 18 months after initial injection
  Objective evaluation of the investigational medical device effect on skin biomechanical properties measurements using Cutometer
Evaluation of product safety | 1 month after each injection for ISRs and 21 months for adverse event collection
  Clinical evaluation of the investigational medical device safety with Injection Site Reactions (ISRs) and adverse event collection

CONTACTS AND LOCATIONS:
Overall Officials: Siham RHARBAOUI, Principal Investigator — Eurofins Laboratoire Dermscan
Locations (1):
- Eurofins Laboratoire Dermscan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No